CLINICAL TRIAL: NCT05831891
Title: A Single-arm, Multicenter, Prospective Clinical Study of Efficacy and Safety of Fruquintinib Combined With Serplulimab in First-line Treatment of Non-clear Renal Cell Carcinoma
Brief Title: Fruquintinib and SeRplulimab: Opening New Frontiers in Treating Non-clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRONTIER
Record Dates: First submitted 2023-04-16; First posted 2023-04-26 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Non-clear Renal Cell Carcinoma
Keywords: Fruquintinib; Serplulimab; combination therapy; first-line; non-clear renal cell carcinoma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Before surgery, patients will receive Fruquintinib 5mg, qd, 2w on/1w off, combined with Serplulimab 4.5mg/kg, IV drip, d1, q3w.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fruquintinib combine with Serplulimab (Experimental): Patients will receive Fruquintinib 5mg, qd, 2w on/1w off, combined with Serplulimab 4.5mg/kg, IV drip, d1, q3w.
  Interventions: Drug: Fruquintinib combined with Serplulimab

INTERVENTIONS:
Drug: Fruquintinib combined with Serplulimab — Fruquintinib 5mg, qd, 2w on/1w off and Serplulimab 4.5mg/kg, IV drip, d1, q3w
  Other Names: Elunate; HLX10

SUMMARY:
This study is design to prospectively investigate the safety and efficacy of Fruquintinib combined with Serplulimab in first-line treatment of non-clear renal cell carcinoma. Fruquintinib, a vascular endothelial growth factor receptor inhibitor, is an anticancer drug independently developed in China to treat refractory metastatic colorectal cancer (mCRC). This is a Single-arm, multicenter, prospective phase 2 clinical study.

DETAILED DESCRIPTION:
The study is ongoing. This is a single-arm, multicenter clinical study enrolling 39 patients with metastatic or unresectable nccRCC at Renji Hospital and Zhongshan Hospital in Shanghai, China. The study is divided into a safety-run-in stage and a cohort expansion stage. Six patients were enrolled in the safety-run-in stage, and no dose-limited toxicity or treatment-related deaths occurred within the 28-day observation period. Consequently, the cohort was expanded to 39 patients. The treatment includes Fruquintinib 5mg, qd, 2w on/1w off, combined with Serplulimab 4.5mg/kg, IV drip, d1, q3w. Tumor response is evaluated at baseline, every 6 weeks during treatment, and at end-of-treatment visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have signed an informed consent form and are willing to complete the study according to the protocol;
2. Age between 18 and 75 years old;
3. Patients with metastatic or unresectable nccRCC who have been histologically or cytologically diagnosed (AJCC 8th edition staging);
4. At least one measurable lesion, as required by the "Measurable Lesion" criteria in RECIST 1.1;
5. Not treated with any systemic anti-tumor therapy since diagnosis, including chemotherapy, targeted therapy, and immunotherapy (including but not limited to anti-PD-1/PD-L1 antibodies, anti-CTLA-4 antibodies, etc.);
6. Expected survival of 3 months;
7. ECOG score 0-1;
8. Good organ function: meeting the following requirements:

   1. Absolute neutrophil count (ANC) ≥1.5× 109/L;
   2. Platelet count ≥100×109/L;
   3. Hemoglobin ≥9g/dL;
   4. Serum albumin ≥2.8g/dL;
   5. Total bilirubin ≤1.5 ×ULN, ALT, AST, and/or ALP ≤3 ×ULN; if liver or bone metastasis is present, ALP ≤5 ×ULN;
   6. Serum creatinine ≤1.5×ULN and creatinine clearance rate 60 mL/min (Cockcroft-Gault, see Appendix 3);
   7. Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤1.5× ULN (patients receiving stable doses of anticoagulant therapy such as low-molecular-weight heparin or warfarin and whose INR is within the expected therapeutic range of anticoagulants can be screened);
9. Patients infected with hepatitis B Virus (HBV) and inactive/asymptomatic carriers, or patients with chronic or active HBV will be allowed to enroll if their HBV DNA<500 IU/mL (or 2500 copies/mL); HCV antibody-positive patients will be allowed to enroll if HCV-RNA is negative during screening.

   Note: HBsAg-positive patients or patients with detectable HBV DNA who receive antiviral treatment should undergo treatment for >2 weeks before enrollment, and continue treatment for 6 months after the study drug treatment.
10. *For women of reproductive age, urine or serum pregnancy test results should be negative within 7 days or less before treatment. And use a medically approved contraceptive (such as an intrauterine device, contraceptive or condom) during the study treatment period and at least 3 months after the last use of Serplulimab and at least 6 months after the last use of chemotherapy;
11. Male subjects who are not sterilized must be willing to use a medically approved contraceptive method (such as an IUD, contraceptive or condom) for the duration of the study treatment, at least 3 months after the last use of Serplulimab and at least 6 months after the last use of chemotherapy.

Exclusion Criteria:

1. There is a history of allergy to any component of the drug SLT or the drug Fruquintinib.
2. A history of or concurrent malignancy (excluding skin basal cell carcinoma and cervical carcinoma in situ and papillary carcinoma of thyroid) that has been cured for more than 5 years and has no active cancer）.
3. Uncontrolled clinical symptoms or diseases of the heart, including: a) NYHA class II or above heart failure; b) unstable angina; c) myocardial infarction within 1 year; d) significant atrial or ventricular arrhythmias requiring clinical intervention.
4. Having received any of the following treatments: a) previous treatment with PD-1, PD-L1 antibodies, or CTLA-4 antibodies; b) received any investigational drugs within 4 weeks prior to the first dose of the study drug; c) enrolled in another clinical trial, unless it is an observational (non-interventional) study; d) requiring systemic treatment with corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive drugs within 2 weeks prior to the first dose of the study drug, with the exception of using corticosteroids for local inflammation or prevention of allergies, nausea, and vomiting. Other special circumstances should be communicated with the investigator. In the absence of active autoimmune diseases, inhaled or locally applied steroids and adrenal cortex hormones that replace a dosage of >10 mg/day prednisone can be used.

   e) Vaccination with anti-tumor vaccines or receipt of live vaccines within 4 weeks prior to the first dose of the study drug; f) underwent major surgery or had any serious trauma within 4 weeks prior to the first dose of the study drug.
5. Toxicity from previous anti-cancer therapy has not recovered to ≤ CTCAE grade 1 (excluding alopecia and residual neurotoxicity related to previous platinum therapy) or does not meet inclusion/exclusion criteria.
6. Serious infection (CTCAE grade >2) within 4 weeks prior to the first dose of the study drug, including severe pneumonia, sepsis requiring hospitalization, and infection-related complications; baseline chest imaging shows active pulmonary inflammation, symptoms and signs of infection within 4 weeks of first dose, or the need for oral or intravenous antibiotics.
7. Active autoimmune diseases or a history of autoimmune diseases (including but not limited to interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism), except autoimmune-mediated hypothyroidism treated with a stable dose of thyroid replacement hormone and I-type diabetes treated with a stable dose of insulin. Patients with vitiligo or childhood asthma/allergy in remission without any intervention in adulthood are not excluded.
8. A history of immunodeficiency diseases, including HIV-positive, other acquired or congenital immunodeficiency diseases, organ transplantation, or allogeneic bone marrow transplantation.
9. A history of interstitial lung disease (excluding radiation pneumonitis that has not been treated with steroids), and a history of non-infectious pneumonia.
10. Evidence of active tuberculosis infection based on medical history and CT examination, a history of active tuberculosis infection within 1 year prior to screening, or a history of active tuberculosis infection over 1 year ago that has not been properly treated.
11. Patients with active hepatitis B (HBV DNA ≥500 IU/mL or 2500 copies/mL) or hepatitis C (positive HCV antibodies and HCV-RNA higher than the detection limit of the assay) are excluded. Patients with HBsAg-positive and HBV DNA-negative or HBV DNA <500 IU/mL or 2500 copies/mL can receive treatment for antiviral therapy for more than 2 weeks before enrolling in the trial and continue antiviral therapy for 6 months after the end of the last dose of the study drug.
12. A known history of psychotropic substance abuse, alcoholism or drug use;
13. Pregnant or lactating women;
14. At the investigator's discretion, patients with other factors that may force them to withdraw from the study, such as concomitant severe illnesses (including mental illness) requiring treatment, significant laboratory abnormalities, and family or social factors that may hinder patient safety or data collection.
15. Patients with severe active bleeding, active peptic ulcers, unhealed gastrointestinal perforations, or gastrointestinal fistulas.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 2 years
  PFS is defined as the time from the the start of treatment till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).

SECONDARY OUTCOMES:
Objective Response Rate | Up to 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1
Disease control rate (DCR) | Up to 2 years
  Disease control rate (DCR) assessed according to RECIST v1.1
Adverse Event | Up to 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0, also types and degree

OTHER OUTCOMES:
Evaluation of potential predictive biomarkers | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No